CLINICAL TRIAL: NCT06428734
Title: Phenotypes, Biomarkers and Pathophysiology in INPH
Brief Title: Clinical Outcome in Patients With INPH
Status: Recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: XWCOPINPH
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Hydrocephalus; Idiopathic Normal Pressure Hydrocephalus; CSF; Glympathic System; Omic
Keywords: Hydrocephalus; Idiopathic Normal Pressure Hydrocephalus
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood, cerebral spinal fluid, saliva, urine, biopsy and autopsy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hydrocephalus: high throughput sequencing and electromyography Whole Genome Sequencing, Whole Exome Sequencing, Transcriptomics, Proteomics, Metabolomics and imaging, such as DTIALPS
  Interventions: Diagnostic Test: hydrocephalus group
- Normal group: Whole Genome Sequencing, Whole Exome Sequencing, Transcriptomics, Proteomics, Metabolomics
  Interventions: Other: normal group

INTERVENTIONS:
Diagnostic Test: hydrocephalus group — Diagnostic Test: high throughput sequencing and electromyography Whole Genome Sequencing, Whole Exome Sequencing, Transcriptomics, Proteomics, Metabolomics and imaging, such as DTIALPS
  Groups: hydrocephalus
Other: normal group — Whole Genome Sequencing, Whole Exome Sequencing, Transcriptomics, Proteomics, Metabolomics and imaging, such as DTIALPS
  Groups: Normal group

SUMMARY:
The aim of this study is to determine the clinical spectrum and natural progression of idiopathic normal pressure hydrocephalus （iNPH ) and related disorders in a prospective single center study, identify digital, imaging and molecular biomarkers that can assist in diagnosis and therapy development and study the etiology and molecular mechanisms of these diseases.

DETAILED DESCRIPTION:
Due to the heterogeneity of the etiology of idiopathic normal pressure hydrocephalus , almost all published studies on the clinical outcome and prognostic factors of iNPH are relatively limited, and most of them are retrospective. It is not clear which is the most reliable predictor of clinical outcome. Therefore, the researchers conducted this prospective cohort study to identify the occurrence, development and outcome of iNPH and determine the main prognostic factors through clinical scales, biomarkers and imaging.

At study visits a standardized clinical examination will be performed including application of clinical rating scales. At all study visits, patients will be asked to donate biosamples; biomaterial collection is optional and participants can elect to participate in sampling of blood, urine, CSF, and/or a muscle biopsy.

Optionally, additional examinations may be performed including imaging，such as DTIALPS, neurophysiological examination, analysis of patient or observer reported outcomes and analysis to characterize molecular biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* patients who was diagnosed as idiopathic normal pressure hydrocephalus

Exclusion Criteria:

* patient received surgical treatment or interventional treatment before patient is pregnant patient unable to complete follow-up patient with other types of hydrocephalus other nervous system diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients who was diagnosed as idiopathic normal pressure hydrocephalus
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
DTIALPS | Change from Baseline at 6 months after VP shunt
  Change of DTIALPS singal intensity in the resting state fMRI in iNPH patients compared with normal healthy group. Also, the responsive and non-responsive iNPH patients functional MRI were analzed.

SECONDARY OUTCOMES:
Kiefer score | Change from Baseline at 6 months after VP shunt
  A score for iNPH severity; range 0-26; higher indicates higher severity.
Mini mental state Examination | Change from Baseline at 6 months after VP shunt
  A score for cognitive ability; range 0-30; higher indicates higher severity.
Gait evaluation | Change from Baseline at 6 months after VP shunt
  10 meters walking test were evaluated of iNPH patients.
modified Rankin scale | Change from Baseline at 6 months after VP shunt
  A score for functional neurological status ; range 0-5; higher indicates higher severity.
Change in the resting state fMRI | Change from Baseline at 6 months after VP shunt
  Change of BOLD singal intensity in the resting state fMRI in iNPH patients compared with normal healthy group. Also, the responsive and non-responsive iNPH patients functional MRI were analzed.
omic pattern of CSF in iNPH patients | Before surgery in lumbar CSF
  Comparing the omic pattern differences in CSF between iNPH patients and normal age-matched normal volunteers by the analysis of mass spectrometry. Also, the responsive and non-responsive iNPH patients omic pattern were analzed.
omic pattern of CSF in iNPH patients | Change from Baseline at 6 months after VP shunt
  Comparing the omic pattern differences in CSF of iNPH patients before surgery and after VP shunt by the analysis of mass spectrometry. Also, the responsive and non-responsive iNPH patients omic pattern were analzed.

CONTACTS AND LOCATIONS:
Locations (1):
- Fengzeng Jian, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Zhang C, Xu K, Zhang H, Sha J, Yang H, Zhao H, Chen N, Li K. Recovery of glymphatic system function in patients with temporal lobe epilepsy after surgery. Eur Radiol. 2023 Sep;33(9):6116-6123. doi: 10.1007/s00330-023-09588-y. Epub 2023 Apr 3. PMID 37010581
- [Background] Georgiopoulos C, Tisell A, Holmgren RT, Eleftheriou A, Rydja J, Lundin F, Tobieson L. Noninvasive assessment of glymphatic dysfunction in idiopathic normal pressure hydrocephalus with diffusion tensor imaging. J Neurosurg. 2023 Sep 8;140(3):612-620. doi: 10.3171/2023.6.JNS23260. Print 2024 Mar 1. PMID 37724800
- [Background] Yuan C, Xia P, Duan W, Wang J, Guan J, Du Y, Zhang C, Liu Z, Wang K, Wang Z, Wang X, Wu H, Chen Z, Jian F. Long-Term Impairment of the Blood-Spinal Cord Barrier in Patients With Post-Traumatic Syringomyelia and its Effect on Prognosis. Spine (Phila Pa 1976). 2024 Mar 15;49(6):E62-E71. doi: 10.1097/BRS.0000000000004884. Epub 2023 Nov 28. PMID 38014747